CLINICAL TRIAL: NCT02349503
Title: A Phase 1, Open-Label, Single-Dose, Sequential Dose-Escalation Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of NBI-77860 in Adolescent Females With Congenital Adrenal Hyperplasia
Brief Title: Safety, Pharmacokinetics and Pharmacodynamics of NBI-77860 in Adolescent Females With Congenital Adrenal Hyperplasia
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Sponsor: Neurocrine Biosciences (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NBI-77860-1401
Record Dates: First submitted 2015-01-20; First posted 2015-01-29 (Estimated); Last update posted 2015-06-11 (Estimated); Status verified 2015-06

CONDITIONS: Congenital Adrenal Hyperplasia
Keywords: Adrenocortical function; Adrenal hyperplasia, Congenital; 21-hydroxylase deficiency; Adrenogenital Syndrome; Adolescents; Female; Hyperplasia; Adrenal Gland Diseases; Congenital Abnormalities; Adrenocortical Hyperfunction; Disorders of Sex Development; Endocrine System Diseases; Genetic Diseases, Inborn; Gonadal Disorders; Metabolic Diseases; Metabolism, Inborn Errors; Pathologic Processes; Steroid Metabolism, Inborn Errors; Urogenital Abnormalities; Corticotropin Releasing Factor
MeSH Terms: conditions — Adrenal Hyperplasia, Congenital; Congenital adrenal hyperplasia due to 21 hydroxylase deficiency; Adrenogenital Syndrome; Hyperplasia; Adrenal Gland Diseases; Congenital Abnormalities; Adrenocortical Hyperfunction; Disorders of Sex Development; Endocrine System Diseases; Genetic Diseases, Inborn; Gonadal Disorders; Metabolic Diseases; Metabolism, Inborn Errors; Pathologic Processes; Steroid Metabolism, Inborn Errors; Urogenital Abnormalities | interventions — NBI 77860

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- NBI-77860 Dose Group1 (Experimental): NBI-77860 administered orally on Night 1 at bedtime (at approximately 2200 hours).
  Interventions: Drug: NBI-77860
- NBI-77860 Dose Group 2 (Experimental): NBI-77860 administered orally on Night 1 at bedtime (at approximately 2200 hours). Dosing will not commence until all safety and PK results from the dose group 1 have been reviewed to ensure there are no safety concerns and that maximum tolerated dose (MTD) has not been reached.
  Interventions: Drug: NBI-77860
- NBI-77860 Dose Group 3 (Experimental): NBI-77860 administered orally on Night 1 at bedtime (at approximately 2200 hours). Dosing will not commence until all safety and PK results from the dose group 2 have been reviewed to ensure there are no safety concerns and that maximum tolerated dose (MTD) has not been reached.
  Interventions: Drug: NBI-77860

INTERVENTIONS:
Drug: NBI-77860
  Arms: NBI-77860 Dose Group1
Drug: NBI-77860
  Arms: NBI-77860 Dose Group 2
Drug: NBI-77860
  Arms: NBI-77860 Dose Group 3

SUMMARY:
This is a Phase 1, multicenter, open-label, single-dose study to evaluate the safety and tolerability, pharmacokinetics (PK), and pharmacodynamics (PD) of NBI-77860 in subjects with congenital adrenal hyperplasia (CAH). The study will be conducted in approximately 15 adolescent females (12-18 years of age) with a documented medical diagnosis of classic 21-hydroxylase deficiency CAH. The study will include three independent dose cohorts of NBI-77860 (approximately 5 subjects per dose cohort). Ascending doses will be evaluated as part of a sequential-cohort design.

ELIGIBILITY:
Inclusion Criteria:

1. Have documentation of written informed consent, or written and witnessed assent from the subject and written informed consent from the subject's parent or legal guardian.
2. Be in good general health.
3. Have a medically confirmed diagnosis of classic 21-hydroxylase deficiency CAH.
4. Be on a stable regimen of steroidal treatment for CAH for a minimum of 30 days before baseline (Night 1) that is expected to remain stable throughout the study.
5. Subjects of childbearing potential must be instructed on the proper use of barrier methods of contraception and agree to use hormonal or two forms of nonhormonal contraception (dual contraception) consistently from screening until the final study visit or 30 days after the last dose of study drug, whichever is longer.
6. Subjects of childbearing potential must have a negative pregnancy test at screening and negative urine pregnancy test at baseline (Night 1).
7. Have a negative urine drug (for illegal drugs) and alcohol breath test at screening and baseline (Night 1).
8. Be willing and able to adhere to the study regimen and study procedures described in the protocol and informed consent/assent form, including all requirements at the study center and return for the follow-up visit.
9. Be willing to provide authorization for access to personal health information in conjunction with US Health Insurance Portability and Accountability Act (HIPAA).

Exclusion Criteria:

1. Have a clinically significant unstable medical condition or chronic disease, or malignancy.
2. Had a medically significant illness within 30 days of screening.
3. Have a known or suspected differential diagnosis of any of the other known forms of classic CAH.
4. Have a history that includes bilateral adrenalectomy, hypopituitarism, or other condition requiring daily therapy with orally administered glucocorticoids.
5. Pregnant or lactating females.
6. Have a history of epilepsy or serious head injury.
7. Test positive at screening for hepatitis B, hepatitis C, or human immunodeficiency virus (HIV), or have a history of a positive result.
8. Have a recent history (≤1 year) of alcohol or drug abuse, or current evidence of substance dependence or abuse criteria.
9. Used any other investigational drug within 30 days before initial screening, or plans to use an investigational drug (other than the study drug) during the study.
10. Have a blood loss ≥250 mL or donated blood within 56 days or donated plasma within 7 days before baseline.
11. Self-report consumption of more than 6 caffeine-containing beverages a day within the last month before baseline.

Ages: 12 Years to 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2015-02; Primary Completion 2015-10 (Estimated); Study Completion 2015-10 (Estimated)

PRIMARY OUTCOMES:
Number of participants with adverse events following one oral dose of NBI-77860 | Up to 8 weeks

SECONDARY OUTCOMES:
Area Under Concentration Curve (AUC) of NBI-77860 and its metabolites following one oral dose of NBI-77860 | Night 1 and Days 2, 7, 14, 21 and 35 (or early termination)
Concentrations of 17-hydroxyprogesterone (17-OHP) following one oral dose of NBI-77860 | Screening, Night 1, Day 2 (10, 12 and 24 hours postdose) and 35 (or early termination)
Concentrations of adrenocorticotropin hormone (ACTH) following one oral dose of NBI-77860 | Screening, Night 1, Day 2 (10, 12 and 24 hours postdose) and 35 (or early termination)

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Ann Arbor, Michigan
  - Seattle, Washington